CLINICAL TRIAL: NCT02816814
Title: Effects of a Lacto-ovo-vegetarian Diet Riched in Omega-3 Fatty Acids on the Lipidomic Membrane Profile of Erythrocyte in Menopausal Women.
Brief Title: Lacto-ovo-vegetarian Diet Riched in Omega-3 Fatty Acids in Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Maria Gabriella Caruso, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RC242016
Record Dates: First submitted 2016-06-17; First posted 2016-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Menopause; Metabolic Syndrome; Hepatic Steatosis
Keywords: Menopause; Diet; Lipidomic profile; Vasomotor symptoms; Omega-3 fatty acids
MeSH Terms: conditions — Metabolic Syndrome; Fatty Liver | interventions — Fatty Acids, Omega-3; Diet

ARMS (2):
- Love Diet (Active Comparator): Overweight females (BMI > 25) in menopause
  Interventions: Other: Diet with extra virgin olive oil
- LωVE diet (Experimental): Overweight females (BMI > 25) in menopause
  Interventions: Other: Diet rich in omega-3 fatty acids

INTERVENTIONS:
Other: Diet rich in omega-3 fatty acids — A diet rich in omega-3 fatty acids (7g/die) will be administered for 4 months to overwieght women in menopause
  Arms: LωVE diet
Other: Diet with extra virgin olive oil — A diet rich in EVO (25-30g/die) will be administered for 4 months to overwieght women in menopause
  Arms: Love Diet

SUMMARY:
Healthy lifestyle, based on healthy diet and exercise, is a key factor to prevent the most common menopausal disorders and chronic diseases to which women are more exposed during this life stage. Therefore, menopausal women may represent a target for evaluating the effectiveness of nutritional intervention studies based on protective diets against the common metabolic diseases, such as metabolic syndrome, obesity and hepatic steatosis.

Lipidomics aims to study the lipid molecules in a "dynamic" way and allows to define not only structure and functions of a set of lipid species present in an organism, but also the changes that occur during cell metabolism under physiological and pathological conditions in order to understand their role as part of the complex functional balance of a living organism.

Quantitative and qualitative determination of fatty acids profiles in cell membranes allows to follow their molecular changes occurring for intrinsic and extrinsic metabolic causes, such as inflammation, stress, nutrition.

Scientific evidence has shown that, for nutritional studies, the most representative cell is the erythrocyte, which is a biomarker of an individual's general state of health. In fact, the evaluation of the fatty acid composition contained in the membrane of red blood cell, which has an half-life of four months, allows to follow the nutritional status of a subject and to acquire information about his eating habits, with special reference to fat consumption.

The higher intake of omega-3 fatty acids is associated with a decreased inflammatory state which is often altered in patients with metabolic diseases, hepatic steatosis and obesity.

Overweight or obese women in menopause for at least 12 months, aged between 45 and 68 years, will be submitted at baseline to blood samples for lipidomic profile, blood tests, medical examination with blood pressure and anthropometric measurements (weight, height, waist and hip circumferences), indirect calorimetry and bioimpedentiometry. Participants will be randomly assigned to diet with extra virgin olive oil (LoVE DIET) or to diet riched in omega-3 fatty acids (LωVE DIET) for four months. During the treatment period, women enrolled will undergo medical examination and dietary control to assess the adherence to the dietary pattern, collecting anthropometric measurements, indirect calorimetry and bioimpedentiometry after 4 and 16 weeks as well as blood samples after 16 weeks.

The results will be analyzed using appropriate statistical tests. All patients will be made to sign an informed consent.

ELIGIBILITY:
Inclusion Criteria will be: post-menopausal female women with BMI 25-33; baseline fasting glucose<110 mg/dl; total cholesterol ranging from 200 mg/dl and 260 mg/dl; triglycerides ranging from150 mg/dl and 200 mg/dl.

Exclusion Criteria will be: hormone replacement therapy, lipid-lowering therapy, use of corticosteroids and/or nutraceutics in the previous six months, patients with a history of cancer or in chemotherapy.

Ages: 45 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Fatty acids quantification by GC and expressed as ppm in erythrocyte membranes | 4 months
  Quantitative analysis of the fatty acids composition of erythrocyte membranes using gas cromatography

SECONDARY OUTCOMES:
Vasomotor menopausal symptoms by Kupermann scale | Baseline, 1 month, 4 months
  Vasomotor menopausal symptoms will be registered using a standardised questionnaire (Kupperman scale

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Specializzata in Gastroenterologia Saverio de Bellis, Castellana Grotte, Bari, Italy